CLINICAL TRIAL: NCT05776810
Title: Syncope Trial to Understand Tilt Testing or ECG Recording. Tenth Prevention of Syncope
Brief Title: Syncope Trial to Understand Tilt Testing or ECG Recording Tenth Prevention of Syncope Trial
Acronym: (POST10)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: POST 10
Record Dates: First submitted 2023-03-01; First posted 2023-03-20 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-05

CONDITIONS: Syncope
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All eligible participants (Experimental): All eligible participants are randomly assigned to one of two interventions- early Head-Up Tilt Table procedure or early Implantable Loop Recorder. The assignment is random and at a 1:1 ratio between the two strategies.
  Interventions:
  Diagnostic Test: Head Up Tilt Table (HUT) Device: Implantable Loop Recorder
  Interventions: Diagnostic Test: Diagnostic Test: Head Up Tilt Table (HUT); Device: Device: Implantable Loop Recorder

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: Head Up Tilt Table (HUT) — Participant randomized to open-label diagnostic strategy. Results and all follow-up care to be in the hands of treating cardiologist as this is a pragmatic study.
  the early HUT [protocol: supine pre-tilt phase 5 min, un-medicated HUT to 70 degrees for 20 minutes; if response negative then 400 μg of sublingual nitroglycerin and continued 70 degree tilt for 20 minutes]
Device: Device: Implantable Loop Recorder — ILR is a small subcutaneously implanted device, lasting up to 3 years, that records heart rhythms, and which may be either auto-triggered or patientactivated.

SUMMARY:
The Study To Understand Tilt Tests versus Extended Recordings (STUTTER, POST 10) will test the hypothesis that first performing a diagnostic HUT in older patients with syncope of unknown cause will provide earlier and more diagnoses than inserting an ICM.

DETAILED DESCRIPTION:
A total of 144 patients ≥50 years old with ≥1 syncopal spell in the preceding year who lack a clear etiologic diagnosis for syncope and no clinically apparent structural heart disease will be randomized to first undergo HUT or to first receive an ICM in an open label, parallel group study. The primary outcome measure will be the establishment of a documented etiologic diagnosis of the cause of syncope, defined below. This will be a formal pragmatic study of two diagnostic strategies, designed around the PRECIS2 criteria. The key question addresses which test should be done first, and beyond that care will be left in the hands of the specialist physician with primary responsibility for assessing and managing syncope.

This is a Pragmatic Trial, which is a rigorous randomized trial method that enables the study of interventions in the real world. Pragmatic trials are designed to determine the effects of an intervention under the usual conditions in which it will be applied, in contrast to conventional explanatory biomedical trials that are designed to determine the effects of an intervention under ideal circumstances. The researcher's touchstone is usual syncope specialist management. There are 9 criteria of the PRECIS2 tool for pragmatic trials:1) similarity of eligibility criteria to usual care, 2) no extra recruitment effort, 3) similar setting to usual care, 4) similar health care organization and delivery to usual care, 5) similar flexibility to usual care, 6) similar flexibility in patient monitoring, 7) similar follow-up intensity to usual care, 8) direct relevance of primary outcome to participants, and 9) completeness of data inclusion. Each criterion is scored 1-5; the researchers provide these scores for each criterion. Study design and conduct are designed to resemble real clinical practice with its variable conduct and decision-making. The primary outcome is establishing a diagnosis by one of two recommended methods, and both methods have evidence-based criteria. the researchers will issue a brochure to remind investigators of the guidelines' criteria. Both have objective ECG criteria and tilt tests have BP criteria. Bias is a concern, and the Outcomes Adjudication Committee will adjudicate post hoc all results blindly.

ELIGIBILITY:
Inclusion Criteria:

* age >50 years old
* ≥1 syncope26 in the prior 12 months
* diagnosis unclear after history, physical exam, and electrocardiogram
* no apparent risk of death due to the cause of syncope

Exclusion Criteria:

* cannot provide informed consent or attend routine follow up
* have known left ventricular ejection fraction < 50%,or have
* pacemaker, ICD, or ICM
* Class I indication for permanent pacing or ICD implantation
* hypertrophic cardiomyopathy
* a history of myocardial infarction within 3 months prior to enrolment
* a major chronic co-morbid medical condition that would preclude 12 months of follow-up
* bifascicular block
* epilepsy proven by electroencephalography
* syncope of known cause

Ages: 50 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be the determination of the diagnosis of the cause of syncope (PRECIS2 criterion 8, 5/5) within 2 years. | within 2 years

SECONDARY OUTCOMES:
cost from the perspective of the health care system | Within 2 years
psychometric quality of life | Within 2 years
sex and gender, and patient preferences. | Within 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Happ S, Raj SR, Chew D, Sheldon R. Physician Perspectives on the Initial Diagnostic Strategy of Syncope in Older Patients Without Diagnostic Clues. Ann Noninvasive Electrocardiol. 2026 Mar;31(2):e70155. doi: 10.1111/anec.70155. PMID 41614589